CLINICAL TRIAL: NCT02012582
Title: An Exploratory Phase 2 a Study to Assess Safety, Tolerability, Pharmacodynamic and Pharmacokinetics of VAS203 in Patients With Moderate and Severe Traumatic Brain Injury
Brief Title: Phase 2 a Study to Assess Safety and Pharmacokinetics of VAS203 in Patients With Traumatic Brain Injury
Acronym: NOSTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: veriNOS operations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAS203/II/1/03
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — 4-amino-tetrahydrobiopterin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VAS203 15 mg/kg (Experimental): Three 5 mg/kg/12-hours infusion with 12 hours break after each infusion. Total dose: 15 mg/kg
  Interventions: Drug: VAS203
- VAS203 20 mg/kg (Experimental): 10 mg/kg/24 hours, 48 hour continuous infusion. Total dose: 20 mg/kg
  Interventions: Drug: VAS203
- VAS203 30 mg/kg (Experimental): 10 mg/kg/24 hours, 72 hour continuous infusion. Total dose: 30 mg/kg
  Interventions: Drug: VAS203
- Saline (Placebo Comparator): 0.9 % Sodium chloride infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: VAS203 — i.v. infusion
  Other Names: Ronopterin
  Arms: VAS203 15 mg/kg; VAS203 20 mg/kg; VAS203 30 mg/kg
Drug: Saline — i.v. infusion
  Other Names: 0.9 % NaCl
  Arms: Saline

SUMMARY:
In the exploratory multi-center Phase 2 a study safety, tolerability, pharmacodynamics and pharmacokinetics of the Nitric Oxide Synthase inhibitor VAS203 is assessed in patients with moderate and severe traumatic brain injury. Traumatic brain injury patients (32 males) receive 15, 20 and 30 mg/kg VAS203, respectively, by continuous infusion in three cohorts (Cohort 1 open; Cohorts 2 and 3 double blind, randomised placebo-controlled). End of Study for all patients will be Day 14; adverse events and concomitant medications will be documented throughout the study.

Objectives are to assess safety and tolerability of VAS203, to evaluate concentrations of metabolites of VAS203 in plasma and microdialysate and to assess pharmacodynamic effects of VAS203 on surrogate parameters. Safety parameter will include vital signs (blood pressure heart rate, respiration rate, oxygen saturation and blood gases), fluid balance, ECG, laboratory examinations (clinical chemistry, liver function, haematology/coagulation, urinalysis, renal parameters) and adverse events. Concentration of VAS203 will be determined in plasma and microdialysate. Pharmacodynamic parameters will include intracranial pressure (ICP), biochemical parameters in microdialysate (nitrite/nitrate, arginine, citrulline, pyruvate, lactate, glucose), Partial Oxygen Pressure in brain parenchyma and Therapy Intensity Level (TIL).

DETAILED DESCRIPTION:
Intravenous administration of study medication for each patient will start as soon as possible but not later than 12 hours after trauma. Patients in Group 1 will receive open label study drug (VAS203). Patients in Group 2 and 3 will be randomised to treatment with VAS203 or placebo.

In addition to study treatment, each patient will receive the best "standard of care" for the study centre; no treatment will be withheld.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patient's legal guardian or legal representative
* 18 - 65 years of age, inclusive
* Head trauma within the last 12 hours
* Traumatic brain injury with Glasgow Coma Score (GCS) ≥ 5 and that requires ICP monitoring
* Catheter placement for monitoring and management of increased ICP
* Microdialysis probe placement in penumbra zone or ipsilateral to contusion if focal
* Systolic blood pressure ≥ 100 mmHg
* Females of child-bearing potential must have a negative pregnancy test

Exclusion Criteria:

* Penetrating head injury (e.g. missile, stab wound)
* Not expected to survive more than 24 hours after admission
* Concurrent, but not pre-existing, spinal cord injury
* Unilateral and bilateral fixed and dilated pupil (> 4 mm)
* Cardiopulmonary resuscitation performed post injury
* continuing bleeding likely to require multiple transfusions (> 4 units red blood cells)
* Coma due to a "pure" epidural hematoma (lucid interval and absence of structural brain damage on CT scan)
* Coma suspected to be primarily due to other causes than head injury (e.g. drug overdose)
* Known or CT scan evidence of pre-existing major cerebral damage
* Decompressive craniectomy, planned prior to randomization
* Polytraumatic patients with Injury Severity Score > 25, or rhabdomyolysis
* Injuries to ascending aorta and/or carotid arteries
* serum creatinine values > 1.5 mg/dL
* estimated Glomerular Filtration Rate < 60 ml/min (MDRD-formula)
* body mass index (BMI) > 35, Body weight > 120 kg
* Any severe concomitant condition (cancer; hematologic, renal, hepatic, coronary disease; major psychiatric disorder; alcohol or drug abuse), that can be ascertained at admission
* Known to have received an experimental drug within 4 weeks prior to current injury
* Administration of > 100 ml of contrast media containing iodine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tegtmeier, Dr., Study Director — veriNOS operations GmbH
Locations (6):
- Medical University Innsbruck Department of Neurology, Innsbruck, Austria
- HIA Sainte-Anne Boulevard Sainte-Anne, Toulon, France
- Spain (2):
  - Vall d'Hebron University Hospital Department of Neurosurgery, Barcelona
  - Hospital Clinic University of Barcelona Surgical Intensive Care Unit, Barcelona
- University Hospital Zuerich Surgical Intensive Care, Zurich, Switzerland
- Southampton University Hospital Division of Clinical Neurosciences, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stover JF, Belli A, Boret H, Bulters D, Sahuquillo J, Schmutzhard E, Zavala E, Ungerstedt U, Schinzel R, Tegtmeier F; NOSTRA Investigators. Nitric oxide synthase inhibition with the antipterin VAS203 improves outcome in moderate and severe traumatic brain injury: a placebo-controlled randomized Phase IIa trial (NOSTRA). J Neurotrauma. 2014 Oct 1;31(19):1599-606. doi: 10.1089/neu.2014.3344. Epub 2014 Jul 28. PMID 24831445

RESULTS

PARTICIPANT FLOW:
Groups:
- VAS203 15 mg/kg: Three 5 mg/kg/12-hours infusion with 12 hours break after each infusion. Total dose: 15 mg/kg
  VAS203
- VAS203 20 mg/kg: 10 mg/kg/24 hours, 48 hour continuous infusion. Total dose: 20 mg/kg
  VAS203
- VAS203 30 mg/kg: 10 mg/kg/24 hours, 72 hour continuous infusion. Total dose: 30 mg/kg
  VAS203
- Placebo: 0.9 % Sodium chloride infusion
  Placebo
Period: Overall Study
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 0.9 % Sodium chloride infusion
  Saline
- Total: Total of all reporting groups
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Full Range); unit: years] | 36.6 [21 to 59] | 34.8 [21 to 61] | 45.3 [31 to 65] | 35.9 [26 to 54] | 38.9 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 2 | 6
  Male | 8 | 5 | 7 | 6 | 26
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 0 | 1 | 1 | 2
  United Kingdom | 2 | 0 | 1 | 0 | 3
  France | 1 | 1 | 1 | 2 | 5
  Switzerland | 1 | 5 | 2 | 1 | 9
  Spain | 4 | 2 | 3 | 4 | 13

OUTCOME MEASURES:

1. Secondary Outcome: Duration (Number of Time-points) of Intracranial Pressure (ICP) > 20 mmHg
Time Frame: Hourly from start of infusion to 144 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 9 (13.3) | 9 (13.8) | 12.9 (29.5) | 12.8 (16.4)

2. Secondary Outcome: Duration (Number of Hours) of Cerebral Perfusion Pressure (CPP) < 60 mmHg
Description: Duration (number of hours) of cerebral perfusion pressure (CPP) < 60 mmHg calculated from ICP and mean arterial blood pressure (MAP): CPP = MAP - ICP)
Time Frame: Hourly from start of infusion to 144 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 16.5 (26.9) | 5.9 (8) | 11.8 (14.4) | 9.4 (9.4)

3. Secondary Outcome: Therapy Intensity Level Score
Description: Therapy Intensity Level Score: Total Score calculated daily as the sum of all individual measures, range from 3 (good outcome) to 50 (worst outcome):
  Scores:
  0-2 Head elevation 0-8 Sedation 0-1 Paralysis 1-3 Hyperventilation 0-2 Increased Oxygenation 1-3 Cooling 0-2 Osmotherapy 0-3 CSF Drainage 0-1 Red Blood Cell Transfusion 1-3 Cerebral perfusion pressure 0-1 Surgery for mass lesion 0/5/10 none/unilateral/bilateral Decompressive Craniectomy 0/10 Laparatomy to treat intracranial hypertension due to abdominal hypertension
Time Frame: Daily from day 1 to day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
units on a scale
  Day 1 | 11.4 (3.5) | 11.8 (3.5) | 10 (2.6) | 11.3 (2.6)
  Day 2 | 11.1 (1.6) | 10.5 (3.7) | 10.3 (3.5) | 11.5 (3.2)
  Day 3 | 10.5 (2) | 9.1 (4.1) | 9.3 (2.6) | 12.3 (5.7)
  Day 4 | 10.4 (3.2) | 9.6 (4.5) | 8.9 (3.3) | 12.4 (6.5)
  Day 5 | 9.6 (3.1) | 9.5 (4.7) | 8.8 (3.5) | 12.7 (5.5)
  Day 6 | 9 (2.8) | 9.5 (4.7) | 8.1 (4.7) | 12 (3.6)
Statistical Analysis 1: Comparison: VAS203 15 mg/kg vs VAS203 20 mg/kg vs VAS203 30 mg/kg vs Placebo; Placebo versus pooled VAS203 Arms/Groups; Test type: Superiority or Other; p < 0.04, Mixed Models Analysis — Mixed model analysis for TIL with the patient as random effect and study day, cohort, treatment, and interaction between study day and treatment as fixed effects

4. Post Hoc Outcome: Extended Glasgow Outcome Score (eGOS)
Description: Scoring: Range from 1 (worst outcome) to 8 (good outcome). The patient´s overall rating is based on the lowest outcome category indicated on the scale.
  Score Description
  1. Dead
  2. Vegetative State
  3. Lower Severe Disability
  4. Upper Severe Disability
  5. Lower Moderate Disability
  6. Upper Moderate Disability
  7. Lower Good Recovery
  8. Upper Good Recovery
Time Frame: 6 months after start of treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
units on a scale | 6.5 [3 to 7] | 7 [4 to 8] | 6 [3 to 7] | 4.5 [1 to 6]
Statistical Analysis 1: Comparison: VAS203 15 mg/kg vs VAS203 20 mg/kg vs VAS203 30 mg/kg vs Placebo; Placebo versus pooled VAS203 Arms/Group; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis

5. Primary Outcome: Safety and Tolerability of VAS203 in Patients With Moderate and Severe TBI
Description: Tolerability (good, satisfactory, sufficient, poor) of VAS203 in patients with moderate and severe TBI, as judged by the investigators at day 14.
  Safety outcome measure description see safety section
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
participants
  Tolerability good | 8 | 8 | 6 | 8
  Tolerability poor | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Daily assessment by investigator
Arm/Group | VAS203 15 mg/kg | VAS203 20 mg/kg | VAS203 30 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 4/8 | 2/8
Other Adverse Events (participants affected / at risk) | 6/8 | 7/8 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAS203 15 mg/kg (N=8) | VAS203 20 mg/kg (N=8) | VAS203 30 mg/kg (N=8) | Placebo (N=8)
Pupils unequal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain death (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAS203 15 mg/kg (N=8) | VAS203 20 mg/kg (N=8) | VAS203 30 mg/kg (N=8) | Placebo (N=8)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 3 (4) | 2 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheder site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Phosphorus decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood uric acid decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CRP increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Urine analysis abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Adrenergic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ICP increase (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No